CLINICAL TRIAL: NCT01414582
Title: Transcranial Direct Current Stimulation (tDCS) as a Potential Adjunct Intervention in Stroke Rehabilitation
Brief Title: Transcranial Stimulation and Motor Training in Stroke Rehabilitation
Acronym: tDCS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); The Dunhill Medical Trust (Other)
Responsible Party: Heather House, University of Oxford Research Services
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10/H0604/98
Record Dates: First submitted 2011-08-04; First posted 2011-08-11 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Stroke; Cerebral Infarction; Cerebrovascular Disorders; Brain Diseases
Keywords: tDCS; Stroke; Functional MRI; Motor Learning
MeSH Terms: conditions — Stroke; Cerebral Infarction; Cerebrovascular Disorders; Brain Diseases | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anodal tDCS and Motor Training (Experimental): Participants will receive anodal tDCS over the primary motor cortex of the ipsilesional hemisphere. The following parameters will be used: stimulation intensity of 1mA for the first 20 minutes of motor training (9 consecutive sessions Monday-Friday).
  Interventions: Device: Anodal tDCS; Other: Motor Training
- Sham tDCS and Motor Training (Sham Comparator): Participants will receive sham tDCS over the primary motor cortex of the ipsilesional hemisphere for the first 20 minutes of motor training (9 consecutive sessions Monday-Friday).
  Interventions: Other: Motor Training

INTERVENTIONS:
Device: Anodal tDCS — Participants will receive anodal tDCS over the primary motor cortex of the ipsilesional hemisphere. The following parameters will be used: stimulation intensity of 1mA for the first 20 minutes of motor training (9 consecutive sessions Monday-Friday).
  Arms: Anodal tDCS and Motor Training
Other: Motor Training — All participants will receive a standardised motor training intervention for the upper paretic limb

SUMMARY:
This study aims to test whether repeated sessions of tDCS result in long-lasting improvements in motor function in patients with chronic stroke.

DETAILED DESCRIPTION:
Previous research that utilises single sessions of tDCS have demonstrated functional improvements; however, these improvements are usually short-lived, lasting less than one hour before the patient's performance returns to baseline. It has been suggested that repeated stimulation sessions are required to elicit long-lasting improvements. We aim to consider these details over the duration of this research, during which patients with chronic stroke will attend for 16 sessions over the course of 3 months.

This research has important implications; previous studies suggest that such an approach has the potential to facilitate physical rehabilitation post-stroke and establish tDCS as a clinically viable rehabilitative tool. Recovery of motor skills may take many months to acquire and therefore strategies that have the potential to enhance acquisition of skill are of practical and scientific interest.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 - 80 years.
* Patients should be at least six months post first symptomatic stroke affecting motor function of the hand.

Exclusion Criteria:

* Anyone who does not have adequate understanding of verbal and written information in English, sufficient to complete any of the safety screening forms.
* Anyone who has a previous history of epilepsy, febrile convulsions as a child or recurrent fainting fits. Likewise, anyone who has a significant family history of epilepsy would be excluded as all these conditions carry a theoretical risk of increasing susceptibility to seizures.
* Any person who has a history of drug abuse or a previous history of a neurological or psychiatric illness, or has a history of neurosurgical procedure is excluded as they may be at increased risk of epilepsy and data collected may be influenced by their condition.
* Patients on some prescription medications such as anti-depressants may be excluded as they may be at an increased risk of seizures.
* Anyone who is currently taking or who has taken anti-malarial treatment in the last 72 hours.
* Pregnant women are excluded as a precaution as there is no data on the effect on maternal cranial stimulation on the fetus.
* Any metallic implant in the neck, head, or eye and anyone with any implanted electrical devices would be excluded as there is a risk of heating with both TMS and TDCS stimulation.
* Anyone with any metal implants or implantable device would be excluded as indicated by the MRI safety screening form. People who suffer with claustrophobia as they are unable to tolerate the scanner.
* Patients who have had more than one stroke. Patients who have had a stroke will also be excluded if they have limited communication in the form of aphasia or a history of dementia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Assessment of Motor Recovery following Stroke | Assessed at 2 separate baseline sessions (at least 1 week apart), and then again immediately following the 9 day intervention (day 10), 1 week, 1 month and 3 months later.
  We are looking for a change in scores between the average of the 2 baseline session scores, and those collected during each follow-up session.
Wolf Motor Function Test | Assessed at 2 separate baseline sessions (at least 1 week apart), and then again immediately following the 9 day intervention (day 10), 1 week, 1 month and 3 months later.
  We are looking for a change in scores between the average of the 2 baseline session scores, and those collected during each follow-up session.
Action Research Arm Test | Assessed at 2 separate baseline sessions (at least 1 week apart), and then again immediately following the 9 day intervention (day 10), 1 week, 1 month and 3 months later.
  We are looking for a change in scores between the average of the 2 baseline session scores, and those collected during each follow-up session.
9 Hole Peg Test | Assessed at 2 separate baseline sessions (at least 1 week apart), and then again immediately following the 9 day intervention (day 10), 1 week, 1 month and 3 months later.
  We are looking for a change in scores between the average of the 2 baseline session scores, and those collected during each follow-up session.

SECONDARY OUTCOMES:
Reaction Time Test | Assessed at 2 separate baseline sessions (at least 1 week apart), and then again immediately following the 9 day intervention (day 10), 1 week, 1 month and 3 months later.
  We are looking for a change in scores between the average of the 2 baseline session scores, and those collected during each follow-up session.
Stroke Impact Scale | Assessed at 2 separate baseline sessions (at least 1 week apart), and then again immediately following the 9 day intervention (day 10), 1 week, 1 month and 3 months later.
  We are looking for a change in scores between the average of the 2 baseline session scores, and those collected during each follow-up session.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Functional MRI of the Brain (FMRIB), Oxford, United Kingdom